CLINICAL TRIAL: NCT01008722
Title: The Dynamics of Human Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sanjiv Narayan, MD, PhD, Professor of Medicine, University of California, San Diego
Other Study IDs: 684; R01HL083359 (NIH)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Atrial Fibrillation; Atrial Tachyarrhythmia
Keywords: Atrial Fibrillation; Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is conducted in patients with atrial fibrillation undergoing clinically prescribed ablation. The study hypothesis is that ablation at specific sites that are identified to 'drive' the atrial fibrillation may improve the success of the ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be patients undergoing electrophysiology study and ablation for paroxysmal or persistent atrial fibrillation (AF) after having failed >or= 1 anti-arrhythmic drug.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be men and women of all races aged 21 to 80 years undergoing clinically indicated ablation of Atrial Fibrillation.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2009-06; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv M. Narayan, MD, PhD, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - University of California, San Diego, La Jolla, California
  - VA San Diego Medical Center, San Diego, California

REFERENCES:
- [Result] Narayan SM, Krummen DE, Shivkumar K, Clopton P, Rappel WJ, Miller JM. Treatment of atrial fibrillation by the ablation of localized sources: CONFIRM (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation) trial. J Am Coll Cardiol. 2012 Aug 14;60(7):628-36. doi: 10.1016/j.jacc.2012.05.022. Epub 2012 Jul 18. PMID 22818076
- [Result] Narayan SM, Krummen DE, Rappel WJ. Clinical mapping approach to diagnose electrical rotors and focal impulse sources for human atrial fibrillation. J Cardiovasc Electrophysiol. 2012 May;23(5):447-54. doi: 10.1111/j.1540-8167.2012.02332.x. Epub 2012 Apr 26. PMID 22537106
- [Result] Narayan SM, Patel J, Mulpuru S, Krummen DE. Focal impulse and rotor modulation ablation of sustaining rotors abruptly terminates persistent atrial fibrillation to sinus rhythm with elimination on follow-up: a video case study. Heart Rhythm. 2012 Sep;9(9):1436-9. doi: 10.1016/j.hrthm.2012.03.055. Epub 2012 Mar 28. No abstract available. PMID 22465458
- [Result] Narayan SM, Krummen DE, Clopton P, Shivkumar K, Miller JM. Direct or coincidental elimination of stable rotors or focal sources may explain successful atrial fibrillation ablation: on-treatment analysis of the CONFIRM trial (Conventional ablation for AF with or without focal impulse and rotor modulation). J Am Coll Cardiol. 2013 Jul 9;62(2):138-147. doi: 10.1016/j.jacc.2013.03.021. Epub 2013 Apr 3. PMID 23563126
- [Result] Narayan SM, Shivkumar K, Krummen DE, Miller JM, Rappel WJ. Panoramic electrophysiological mapping but not electrogram morphology identifies stable sources for human atrial fibrillation: stable atrial fibrillation rotors and focal sources relate poorly to fractionated electrograms. Circ Arrhythm Electrophysiol. 2013 Feb;6(1):58-67. doi: 10.1161/CIRCEP.111.977264. Epub 2013 Feb 7. PMID 23392583
- [Result] Narayan SM, Baykaner T, Clopton P, Schricker A, Lalani GG, Krummen DE, Shivkumar K, Miller JM. Ablation of rotor and focal sources reduces late recurrence of atrial fibrillation compared with trigger ablation alone: extended follow-up of the CONFIRM trial (Conventional Ablation for Atrial Fibrillation With or Without Focal Impulse and Rotor Modulation). J Am Coll Cardiol. 2014 May 6;63(17):1761-8. doi: 10.1016/j.jacc.2014.02.543. Epub 2014 Mar 13. PMID 24632280

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from medical clinic.
Pre-assignment Details: Recruitment from medical clinic.
Groups:
- FIRM-Guided: Consecutive cases of patients undergoing Focal Impulse and Rotor Modulation ablation in addition to Conventional Pulmonary vein isolation (PVI)
- CONVENTIONAL: Consecutive cases of patients undergoing Conventional Pulmonary vein isolation (PVI), but being mapped (Focal Impulse and Rotor Mapping) with basket catheters to identify localized rotational or focal sources. FIRM mapping is performed before ablation, but analysis of maps are performed post-hoc and PVI is blinded to the results from FIRM mapping.
Period: Overall Study
Arm/Group | FIRM-Guided | CONVENTIONAL
Started | 36 (Based on Power Calculations to see 20% outcome improvement by adding FIRM-guided ablation to PVI) | 71 (Based on Power Calculations to see 20% outcome improvement by adding FIRM-guided ablation to PVI)
Completed | 36 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: From Medical Record
Groups:
- Total: Total of all reporting groups
Arm/Group | FIRM-Guided | CONVENTIONAL | Total
Number analyzed (Participants) | 36 | 71 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 55 | 79
  >=65 years | 12 | 16 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9) | 61 (8) | 62 (8)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 34 | 68 | 102
Region of Enrollment [Number; unit: participants]
  United States | 36 | 71 | 107

OUTCOME MEASURES:

1. Primary Outcome: Survival Free of Atrial Fibrillation
Description: Using data from cardiac implanted devices when possible, with recurrence defined as 1% recurrence, or data from intermittent 24-72 hour ambulatory ECGs, with recurrence defined as >30 seconds.
Time Frame: 6 -12 months
Measure: Number; unit: participants
Arm/Group | FIRM-Guided | CONVENTIONAL
Number analyzed (Participants) | 34 | 69
participants | 28 | 31

2. Secondary Outcome: Termination or Slowing of Atrial Fibrillation During Ablation
Description: Using data from electrophysiological study, to determine termination of AF into sinus rhythm or organized atrial tachycardia. or slowing by 10% in cycle length measured on the coronary sinus.
Time Frame: acute
Measure: Count of Participants; unit: Participants
Arm/Group | FIRM-Guided | CONVENTIONAL
Number analyzed (Participants) | 36 | 65
Participants | 31 | 13

ADVERSE EVENTS:
Arm/Group | FIRM-Guided | CONVENTIONAL
Serious Adverse Events (participants affected / at risk) | 2/36 | 6/71
Other Adverse Events (participants affected / at risk) | 0/36 | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FIRM-Guided (N=36) | CONVENTIONAL (N=71)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 2 (2) — Blood in pericardium causing hemodynamic compromise, that requires drainage.
Groin bleed requiring transfusion (Blood and lymphatic system disorders) | 1 (1) | 3 (3) — Groin bleed requiring transfusion
Symptomatic Pulmonary Vein Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Symptomatic Pulmonary Vein Stenosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No